CLINICAL TRIAL: NCT06112210
Title: Effect of Hyperbaric Oxygen Therapy Has no Acute Effects on Recovery and Performance After a Football Match
Brief Title: Effect of Hyperbaric Oxygen Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBstudy
Record Dates: First submitted 2023-10-18; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Performance Enhancing Product Use; Physical Fitness; Recovery; Sport
Keywords: hyperbaric chamber; football; recovery; hyperbaric oxygen therapy; performance; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT group (Experimental)
  Interventions: Other: HBOT group
- CON group (Placebo Comparator)
  Interventions: Other: CON group

INTERVENTIONS:
Other: HBOT group — The HBOT will be performed in a Barox HBOT chamber (Yaklasim Makina San. Ve Tic. Ltd. Sti). Participants will be taken to the chamber immediately after the football match, where they will sit in individual chairs, and oxygen will be delivered through individual masks. The HBOT group will be exposed to 100% oxygen at 2.2 ATA (atmospheres absolute). Session will last 70 minutes.
  Arms: HBOT group
Other: CON group — The placebo protocols will be performed in a Barox HBOT chamber (Yaklasim Makina San. Ve Tic. Ltd. Sti). Participants will be taken to the chamber immediately after the football match, where they will sit in individual chairs, and oxygen will be delivered through individual masks. The CON group will be exposed to normobaric ambient pressure (1 ATA). The session will last 70 minutes.
  Other Names: Control; Placebo
  Arms: CON group

SUMMARY:
The goal of this tudy will be to investigate the effects of a single session of hyperbaric oxygen therapy (HBOT) on recovery and performance after a football match in elite youth football players.

The main questions this study will aim to answer are:

Will a single session of HBOT improve recovery parameters such as biochemical markers and physical fitness in elite youth football players after a football match? Will a single session of HBOT enhance the performance of elite youth football players after a football match?

Participants in this study will include twenty elite youth male football players. They will be randomly assigned to either the HBOT group or the control group. All participants will undergo evaluations for biochemical parameters, physical fitness tests, and the Hooper Index (HI) at multiple time points: before the match, at the end of the match, one hour after the HBOT session, and 12 hours after the HBOT session.

In the HBOT group, participants will receive 100% oxygen under elevated pressure in a hyperbaric chamber for a duration of 70 minutes immediately after the football match. Meanwhile, the control group will be exposed to normal atmospheric pressure.

Biochemical analysis will involve collecting blood samples to measure markers such as myoglobin, creatine kinase, lactate dehydrogenase, alanine aminotransferase, and aspartate aminotransferase. Physical fitness tests will include vertical jump height measurements (squat jump, countermovement jump, and countermovement jump with arm swing) and linear speed assessments at various distances (5 m, 10 m, and 20 m). The Hooper Index (HI) will be used for subjective assessment of fatigue and well-being.

This study aims to provide insights into the potential benefits of HBOT as a recovery strategy for elite youth football players and its impact on performance in the future.

ELIGIBILITY:
Inclusion Criteria:

* football player
* free of injuries
* free of medical conditions contraindicated by hyperbaric oxygen therapy (HBOT)
* written parental consent

Exclusion Criteria:

* pre-existing injuries or medical conditions that are contraindicated by hyperbaric oxygen therapy (HBOT)
* participation in severe physical activity within 24 hours before the study
* participants who do not comply with the requirement to abstain from breakfast, caffeine, and alcohol prior to the first blood collection
* an active respiratory illness, such as a cold, at the time of the study

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Myoglobin | baseline, 3 hours, 5 hours, 24 hours
  Measure of myoglobin concentration in blood. Myoglobin will be determined using Siemens IMMULITE 1000 (Siemens Healthcare Diagnostics, UK).
Creatine kinase | baseline, 3 hours, 5 hours, 24 hours
  Measure of creatine kinase concentration in blood. It will be analyzed using a biochemistry analyzer (A25 Biosystems Chemistry Analyzer).
Lactate dehydrogenase | baseline, 3 hours, 5 hours, 24 hours
  Measure of lactate dehydrogenase concentration in blood. It will be analyzed using a biochemistry analyzer (A25 Biosystems Chemistry Analyzer).
Alanine aminotransferase | baseline, 3 hours, 5 hours, 24 hours
  Measure of alanine aminotransferase concentration in blood. It will be analyzed using a biochemistry analyzer (A25 Biosystems Chemistry Analyzer).
Aspartate aminotransferase | baseline, 3 hours, 5 hours, 24 hours
  Measure of aspartate aminotransferase concentration in blood. It will be analyzed using a biochemistry analyzer (A25 Biosystems Chemistry Analyzer).

SECONDARY OUTCOMES:
Squat jump | baseline, 3 hours, 5 hours, 24 hours
  Measure of a squat jump height in cm. The squat jump will be performed in a semi-squat position with the knees bent at 90 degrees and the arms resting on the hips. Participants will hold this stance for one to three seconds before executing a maximal vertical jump.
Countermovement jump | baseline, 3 hours, 5 hours, 24 hours
  Measure of a countermovement jump height in cm. It will be evaluated with participants standing straight up, distributing their weight equally over both feet. The arms will be secured to the hips to prevent their influence on jump height. Participants will then squat down to a 90-degree flexion and execute a maximal vertical jump without pausing during the change of direction.
Countermovement jump with arm swing | baseline, 3 hours, 5 hours, 24 hours
  Measure of a countermovement jump with arm swing height in cm. It will be evaluated with participants standing straight up, distributing their weight equally over both feet. During the jump, participants will have the freedom to move their arms.
5 meter linear speed | baseline, 3 hours, 5 hours, 24 hours
  Measure of 5 meter linear speed. The Witty photocell system (Witty, System, Microgate, Bolzano, Italy) will be utilized to evaluate performance. These photocells will be positioned 0.4 meters above the ground and will provide measurements with an accuracy of 0.001 meters per second.
10 meter linear speed | baseline, 3 hours, 5 hours, 24 hours
  Measure of 10 meter linear speed. The Witty photocell system (Witty, System, Microgate, Bolzano, Italy) will be utilized to evaluate performance. These photocells will be positioned 0.4 meters above the ground and will provide measurements with an accuracy of 0.001 meters per second.
20 meter linear speed | baseline, 3 hours, 5 hours, 24 hours
  Measure of 20 meter linear speed. The Witty photocell system (Witty, System, Microgate, Bolzano, Italy) will be utilized to evaluate performance. These photocells will be positioned 0.4 meters above the ground and will provide measurements with an accuracy of 0.001 meters per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Hyperbaric center Subotica, Subotica, Serbia